CLINICAL TRIAL: NCT04595214
Title: Develop a Multi-disciplinary Approach for a Personalized Prenatal Diagnostics and Care for Twin Pregnancies
Acronym: PRETWINSCREN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Prof. Ron Maymon, MD, PhD Chairman ObGyn, Assaf-Harofeh Medical Center
Other Study IDs: 0043-20-ASF; JTC 2019-061 2019-00 (Other Grant/Funding Number: ERAPERMED)
Record Dates: First submitted 2020-08-03; First posted 2020-10-20 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Prenatal Disorder; Premature Birth; Twin Pregnancy With Antenatal Problem; Twin; Pregnancy, Affecting Fetus or Newborn; Twin Pregnancy, Antepartum Condition or Complication; Twin Dichorionic Diamniotic Placenta; Twin Monochorionic Monoamniotic Placenta
Keywords: Twin pregnancy; Risk stratification algorithm,; Feto-Maternal complications (preeclampsia, IUGR, PTD, GDM),; TTTS; cfDNA, NIPT
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia; Fetal Growth Retardation | interventions — Divorce

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum and plasma samples are collected at 11-13, 20-22 and 32-34 weeks. Some tested at blood drawing and some are stored at -70oC for testing at study conclusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TTTS cases are treated by intra-uterine laser for separation. — MC twin anaestemosis separatio by laser. Vasa previa and placenta accreta are treated with steroids or other protocols, Positive trisomies by NIPS undergoes CVS or amniocentesis
  Other Names: Placenta previa and acreta are treated according to protocol.; NIPS is used to screen for trisomy 21,13 and 18

SUMMARY:
Different screening modalities evaluation to develop algorithms to predict pregnancy complications in twin pregnancies, and evaluation of serologic response to BNT162b2 Pfeizer/BioNTech vaccination.

DETAILED DESCRIPTION:
This is a multi-center study to identify biomarkers or marker combinations for early prediction of pregnancy complications in twin pregnancies in the first, second or third trimester.

In the future, the identified patients' risk will enable patients' referrals for proper prevention when such will become available

Specifically the investigators aim for

* Predicting the risk to develop preeclampsia, IUGR, preterm delivery, gestational Diabetes Melitus
* Assessment of major and minor markers for chromosomal and structural anomalies
* Identification of placenta accrete spectrum disorders and vasa previa
* Diagnosis of specific MC twin complications such as TTTS

The investigators will stratify and assess all the above according to chorionicity and delivery with complications at <32 weeks, <34 weeks, <37 weeks, and at any gestation.

Screening methods will be conducted in the first, second or third trimester or at any gestation

Also the investigators aim to Identify the risk to lose one or both twins at <32 weeks, <34 weeks, <37 weeks and at any gestation, the ability to predict fetal birth weight at <32 weeks, <34 weeks, <37 weeks and at any gestation

The investigators also aim for monitoring any of the following maternal complications including placental abruption (clinically or on placental examination), postpartum hemorrhage (defined as blood loss ≥1 L within the first 24 hours after birth) at <32 weeks, <34 weeks, <37 weeks and at any gestation.

The investigators will monitor

1. Neonatal morbidity due to intraventricular hemorrhage (IVH) grade II or above - Defined as bleeding into the ventricles, Grade II (moderate) - IVH occupies <50% of the lateral ventricle volume, Grade III (severe) - IVH occupies ≥50% of the lateral ventricle volume or Grade IV (severe) - Hemorrhagic infarction in periventricular white matter ipsilateral to a large IVH
2. Neonatal sepsis confirmed bacteremia in cultures, anemia defined as low Hemoglobin and / or hematocrit requiring blood transfusion, respiratory distress syndrome defined as need for treatment by surfactant and ventilation, necrotizing enterocolitis requiring surgical intervention, and composite of any of the above
3. Newborn admission to neonatal intensive care units (NICU), length of stay and therapies during the admission.
4. Ventilation defined as a need for a positive pressure (continuous positive airway pressure (CPAP), nasal continuous positive airway pressure (NCPAP)) or intubation and a composite of any of the above
5. Any maternal complications within the first 6-10 weeks post delivery. The investigators will recruit patients in the different sites aiming for 1200 twin pregnancy and will collect the patients' entire pregnancy data for developing an algorithm to calculate the risk to develop the complications
6. Evaluation of serologic response to BNT162b2 Pfeizer/BioNTech vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Di-chorionic (DC)or Mono-chorionic (MC) twin pregnancies;
* Both live fetuses at 11+0-13+6 weeks of gestation;
* Informed and written consent

Exclusion Criteria:

* Monoamniotic twins
* Triplet pregnancies that had undergone embryo reduction to twins or with one vanishing twin
* Women who are unconscious or severely ill, those with learning difficulties, or serious mental illness;
* Any other reason the clinical investigators think will prevent the potential participant from complying with the trial protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women with live twin pregnancy at gestational week 11+0 days and 13+6 days
Study Population: This is prospective multi-centre study that includes a site in Israel, two sites in Germany, a site in Catalonia, Spain, a site in Quebec, Canada and a site in the UK. In the participating centres, all eligible women with DC or MC twin pregnancy attending for their routine first hospital visit in pregnancy at 11-13 weeks' gestation will be invited to participate in the trial. pregnancy characteristics will be followed and biomarkers determined. We follow ISUOG and FMF guidelines on how to undertake the appropriate measurements
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | through study completion, an average of 1 year
  preterm delivery before 37 weeks of gestation , or hypertension of >90/140, from gestational week 24 and above throughout pregnancy , baby birth weight below the 5 lower centile for the gestation week, or shoulder dyctorcia at delivery, or newborn admission to NICU for any complication or placental position complications such as placenta accreta, or vasa previa, or intra uterine fetal death,
Adverse neonatal outcome | through study completion, an average of 2 year
  Admission to neonatal intensive care unit, Sepsis, asphyxia, intraventricular hemorrhage, intrauterine growth retardation
Evaluation of serologic response to BNT162b2 Pfeizer/BioNTech vaccination. | through study completion, an average of 2 year including stored samples collected before vaccination was avaluable.
  Testing blood sample drawn for the study for antybody levels in conjunction to BNT162b2 Pfeizer/BioNTech vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ron Maymon, MD,PhD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (7):
- CHU Brugmann,, Brussels, Belgium
- University of Montreal Medical Centre, Canada, Montreal, Canada
- Germany (2):
  - University Hospital Bonn, Bonn, Germany, Bonn
  - Oliver Kagan, Tübingen
- Department of ObGyn, Assaf Harofe-Shamir Medical Center, Zrifin, Israel
- Hospital Clinic, Barcelona,, Barcelona, Catalonia, Spain
- The Fetal Medicine Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
A single database will be unified from all sites. Patents are entered after coding and personal anonymization. Level of sharing will be decided upon the policy of peer review journal. If acessible - dat be stored at the fetal medicine foundation website

REFERENCES:
- [Derived] Svirsky R, Rabbi ML, Hamad RA, Sharabi-Nov A, Kugler N, Galoyan N, Sharon NZ, Meiri H, Maymon R, Levtzion-Korach O. Vaccination in twin pregnancies: comparison between immunization before conception and during pregnancy. Sci Rep. 2024 May 11;14(1):10813. doi: 10.1038/s41598-024-61504-6. PMID 38734805